CLINICAL TRIAL: NCT06381427
Title: Perioperative Interdisciplinary, Intersectoral Process Optimization in Heart Failure: A Multicenter, Prospective-randomized Intervention Study
Brief Title: Perioperative Interdisciplinary, Intersectoral Process Optimization in Heart Failure
Acronym: PeriOP-CARE HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Deutsche Luft und Raumfahrt (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01NVF22109
Record Dates: First submitted 2024-02-26; First posted 2024-04-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Perioperative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): In this group, the anesthesiological risk evaluation is generally conducted in accordance with the current guidelines. Possible additional (instrumental) examinations, intraoperative anesthesiological management, and postoperative inpatient therapy are carried out according to current guidelines and are unaffected by study participation. If services are provided in the control group within the local standards that are also part of the new care model, these will be documented to ensure comparability.
- Intervention group (Active Comparator): A cardiology consultation is conducted, which includes a standardized evaluation. This includes, medical history and physical examination:ECG, Echocardiography, Determination of cardiac troponins and natriuretic peptides in the local central laboratory. The echocardiography aims to qualitatively and quantitatively describe the left and right ventricular systolic and diastolic dimensions and function, as well as the valvular apparatus, the collected findings are presented at the interdisciplinary and intersectoral preoperative medical (POM) conference. Bedside visits with the patient are also possible.During this conference, structured preoperative interdisciplinary and intersectoral case discussions take place, involving the attending outpatient physicians. The POM conference consists of Anesthesiology, Cardiologist, Treating surgeon and optimize preoperative therapy and plan further pre-, intra-, and postoperative as well as outpatient care.
  Interventions: Other: Interdisciplinary decision-making for perioperative care

INTERVENTIONS:
Other: Interdisciplinary decision-making for perioperative care — Interdisciplinary decision-making for perioperative care involving a cardiologist, anesthesiologist, and surgeon in collaboration with the primary care physician. Decisions include determining whether surgery is feasible or if patient optimization is necessary first. Subsequently, targeted postoperative visits by a heart failure nurse and appropriate postoperative care, also after discharge from the hospital, through the primary care physician.
  Arms: Intervention group

SUMMARY:
Chronic heart failure affects up to three million people in Germany, with prevalence increasing with age. It is a leading cause of cardiovascular disease-related deaths. Patients with heart failure undergoing non-cardiac surgery face higher risks of complications and death compared to those with coronary artery disease. Despite guidelines recommending comprehensive preoperative evaluation, there is no systematic risk assessment structure in place, leading to inadequate perioperative care. This study aims to evaluate a multidisciplinary approach for high-risk patients aged 65 and above, regardless of prior heart failure diagnosis, to mitigate postoperative complications. The investigators measure the NTpro BNP before surgery and include patients with NTproBNP> 450 in this study and randomize them either to the standard care group or the intervention group.The hypothesis is that standardized risk screening and multidimensional care (Intervention group) can reduce complications in these patients undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Currently, up to three million people in Germany suffer from chronic heart failure, with prevalence increasing with age. Chronic heart failure ranks among the most common cardiovascular diseases, leading to over 50,000 deaths annually. The proportion of older patients at risk of developing or already having heart failure undergoing non-cardiac surgical procedures is also rising. Studies from the USA indicate that patients with chronic heart failure face a higher risk of cardiac complications, including death, following non-cardiac surgeries compared to those with coronary heart disease. A significant proportion of deaths after non-cardiac surgeries are due to cardiac complications. In Europe, this translates to at least 167,000 cardiac complications annually from non-cardiac surgeries, with around 19,000 being life-threatening. Recent analysis suggests that preoperative elevation of NT-proBNP, a heart failure biomarker, is associated with a significantly increased risk of cardiac complications post-surgery. While German data on this topic are lacking, anesthesia and cardiology guidelines advocate for comprehensive evaluation and risk assessment of heart failure patients before non-cardiac surgeries with medium to high operative risk. However, there's a lack of systematic structures for assessing postoperative morbidity and mortality risks in an interdisciplinary and intersectoral context. Due to workload and resource constraints, comprehensive risk assessments are often delayed until shortly before surgery, leading to inadequate peri- and postoperative care. Evidence supporting improved outcomes through preoperative optimization of heart failure patients and risk-adapted precision medicine for non-cardiac surgeries is also lacking. Consequently, this study aims to evaluate a care model providing multimodal, interdisciplinary, and intersectoral optimization for high-risk patients aged 65 and above with elevated heart failure biomarkers (NT-proBNP>450), regardless of prior heart failure diagnosis. The null hypothesis posits that standardized risk screening and multidimensional interdisciplinary care cannot reduce postoperative complications in these high-risk patients undergoing non-cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Elective non-cardiac surgical operation with intermediate or high operative risk under general anesthesia or combined anesthesia (general and regional anesthesia) as per Figure 1
* ASA (American Society of Anesthesiologists) grade ≥ II
* Qualification for randomization: NT-proBNP ≥ 450pg/ml during routine preoperative evaluation and anesthesia consultation.

Exclusion Criteria:

* Age < 65 years
* Cardiac surgery and cardiology interventional procedures
* Transplantation surgery (e.g., kidney, liver, lung transplantation)
* Kidney surgery (e.g., nephrectomy, partial nephrectomy)
* Procedures involving cardiopulmonary bypass
* Emergency surgery
* Surgery under general anesthesia within the last 30 days
* Primary use of local or regional anesthesia
* Chronic kidney insufficiency with eGFR < 15 ml/min or dialysis-dependent kidney insufficiency
* Surgical time < 30 minutes
* Participation in another interventional study
* Lack of consent
* Limited language proficiency
* Patient's limited or absent capacity to provide consent, as well as patients under legal guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1057 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
combined primary endpoint at 90 days post-operation : re-hospitalization,AKI, bacterial infection and cardiac decompensation | 90 days post-operation
  The combined primary endpoint at 90 days post-operation consists of re-hospitalization for any reason, acute kidney injury according to KDIGO definition, any bacterial infection, and cardiac decompensation.

SECONDARY OUTCOMES:
Incidence of acute kidney injury | at 30 and 90 days
  Indicidence of acute kidney injury based on KDIGO classification, Stage 1,2,3
Incidence of any, treatable, suspected, or confirmed bacterial infection | at 30 and 90 days
  Incidence of any, treatable, suspected, or confirmed bacterial infection
Incidence of cardiac decompensation | at 30 and 90 days
  Incidence of cardiacx decompensation including lung edema, peropheral edema, dyspnoe, pleural effusion
Incidence of re-hospitalization | at 30 and 90 days
  Incidence of re-hospitalization
Mortality | at 30 and 90 days
  Mortality
Incidence of myocardial infarction (STEMI, NSTEMI) | at 30 and 90 days
  Incidence of myocardial infarction (STEMI, NSTEMI)
Incidence of Myocardial Injury after Non-Cardiac Surgery (MINS) | at 30 and 90 days
  Incidence of Myocardial Injury after Non-Cardiac Surgery defined as an elevated troponin level
Quality of life assessed using PHQ-9 | at 30 and 90 days
  Quality of life assessed using Patient Health Questionnaire 9 (PHQ-9), score between 0 and 27, best score is 0
Quality of life assessed using GAD-7 | at 30 and 90 days
  Quality of life assessed using Generalized Anxiety Disorder Scale-7 (GAD-7), score between 0 and 21, best score is 0

OTHER OUTCOMES:
Utilization of services and costs | during the intervention at the hospital
  Utilization of services and costs of each patient during the hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Justus Liebig University Giessen, University Hospital Giessen and Marburg, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] PeriOP-CARE HF study group. Perioperative interdisciplinary optimisation of patients with heart failure undergoing non-cardiac surgery with intermediate or high surgical risk: the rationale and study protocol for the multicentre, randomised interventional PeriOP-CARE HF trial. Clin Res Cardiol. 2025 May;114(5):523-531. doi: 10.1007/s00392-025-02626-3. Epub 2025 Apr 29. PMID 40299034